CLINICAL TRIAL: NCT03280810
Title: Effects of a Psycho-corporal Training on Postural and Cognitive Dual-task Performances in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1708158
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Postural; Cognitive; task
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Movement group (Experimental): patients with schizophrenia (experimental group) have psycho-corporal training once a week, during 1 hour and a half for a period of two months
  Interventions: Other: Movement group
- Control group (No Intervention): No intervervention : patients with schizophrenia (comparator group) who don't have psycho-corporal training

INTERVENTIONS:
Other: Movement group — Experimental group : patients with schizophrenia who realise psycho-corporal training once a week, during 1 hour and a half for a period of two months
  Arms: Movement group

SUMMARY:
Beside these well-known symptoms (positive symptoms (such as delirium and delusions), negative symptoms (such as affective flattening and impoverishment of speech), disorganized behavior, patients with schizophrenia show different kinds of cognitive alterations and motor abnormalities. In schizophrenia, postural impairment could increase the attentional cost of daily motor tasks, leading to a lack of attentional resources, essential to achieve complex cognitive tasks. The intrication of cognitive and postural processings (both impaired in schizophrenia) can be explored by using of a dual-task paradigm.

DETAILED DESCRIPTION:
This study assesses a psycho-corporal training (8 weeks psycho-corporal training) benefits on both postural (increased automation of balance control) and cognitive processings (smaller impact of the dual-task condition on attentional performances) in population of patients suffering from schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* a DSM-IV (Diagnostic and Statistical Manual of Mental Disorders) diagnosis of schizophrenia (men or women)
* Men or woman aged 18-55
* Patients with no change in antipsychotic medication and clinical status within four weeks prior to the study
* Affiliates or entitled to a social security scheme
* Have given their informed consent before participating in the study.

Exclusion Criteria:

* Intelligence Quotient below 70 (score PM38)
* History of head trauma, neurological disease or not stabilized serious physical illness
* Disorders related to the use of a psychoactive substance, as defined by the DSM-IV (abuse, dependence or withdrawal) within 6 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
the losses of postural and attentional control | At 8 weeks
  To analyze the losses of postural and attentional control under dual-task condition.
  Losses of postural and attentional control are calculated by one composite score named mu (Baddeley, Della Sala, Papagno, & Spinnler, 1997).

SECONDARY OUTCOMES:
cognitive decrement | At 8 weeks
  To compare mean values of the cognitive decrement between baseline and 8 weeks in which the Redundancy value of the responses sequence to the random number generation task were analyzed using RgCalc® software (Towse & Neil, 1998).
postural decrement | At 8 weeks
  To compare mean values of the postural decrement between baseline and 8 weeks in which the confidence Ellipse is used as main criteria to evaluate the participants balance ability postural sway platform (WIN-POSTURO Médicapteurs®).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine MASSOUBRE, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No